CLINICAL TRIAL: NCT06369831
Title: Evaluating the Diagnostic Performance of Human Epidermal Growth Factor Receptor 2 (HER2) Targeted Positron Emission Tomography and Computed Tomography (PET/CT) With 68Ga-ABS011 in Metastatic Breast Cancer (mBC)
Brief Title: HER2 Targeted Molecular Imaging in mBC Using 68Ga-ABS011
Acronym: HERMIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abscint NV/SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABS011-1; 2024-511419-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Breast Cancer
Keywords: radiolabeled; single domain antibody; 68Ga; Gallium-68; HER2; PET/CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional, Phase IIb, prospective, single arm radio-diagnostic study.
  Driven by number of biopsied lesions (and not by number of patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-ABS011 PET/CT (Experimental): All Hormone receptor positive/HER2 negative, triple-negative or HER2 positive metastatic Breast Cancer (mBC) patients will undergo a HER2 targeted PET/CT using 68Ga-ABS011 after completion of a 18F-FDG PET/CT and lesion biopsy (and IHC/ISH analysis).
  Interventions: Diagnostic Test: 68Ga-NOTA-ABSCINT-HER2 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-NOTA-ABSCINT-HER2 PET/CT — 68Ga-ABS011, is a single domain antibody (sdAb) with the capability to bind HER2 tumor antigens very fast, while the unbound fraction is rapidly cleared from the blood. ABS011 is labeled with gallium-68, a short-lived isotope (68Ga, t1/2: 68 min). Combining rapid targeting of HER2, fast clearance and low radiation burden make 68Ga-ABS011 is suited for specific tumor marker whole body PET/CT imaging.

SUMMARY:
This phase II study aims to confirm the diagnostic performance and accuracy of 68Ga-ABS011 PET/CT in determining the HER2 expression status, and to evaluate 68Ga-ABS011's ability to drive changes in therapeutic treatment. 68Ga-ABS011 will be compared to the current standard of care (SOCa) diagnostic methods including immunohistochemistry (IHC), in situ hybridization (ISH) and imaging tools used for treatment response follow-up including Fluorodeoxyglucose F-18 (18F-FDG) positron emitted tomography (PET) and contrast enhanced computed tomography (ceCT).

DETAILED DESCRIPTION:
Lesion sampling error resulting tumor heterogeneity is probably the biggest pitfall when determining the HER2 status. Moreover, IHC expression or gene amplification can be affected by procedural differences and sample handling differences that are influenced by the experience and training of the pathologist's team. Last but not least, immunohistochemistry interpretation remains a semiquantitative subjective scoring which is susceptible to considerable interobserver variability.

68Ga-ABS011, is a NOTA (chelating agent to label sdAbs with radionuclides) linked single domain antibody (sdAb) with the capability to bind HER2 tumor antigens very fast, while the unbound fraction is rapidly cleared from the blood. ABS011 is labeled with gallium-68, a short-lived isotope (68Ga, t1/2: 68 min). Combining rapid targeting of HER2, fast clearance and low radiation burden make 68Ga-ABS011 is suited for specific tumor marker whole body PET/CT imaging. The available preclinical and clinical results with 68Ga-ABS011 (or its first generation product), including a phase I and a phase II clinical trials, did not reveal any safety signals. Extended safety assessments, including anti-drug antibody (ADA) serum evaluations after 2 consecutive administrations, supported the previously observed low immunogenicity risk profile with these sdAbs. Besides safety, this tracer showed potential in the assessment of inter-lesional HER2 expression heterogeneity and also displayed some higher sensitive and more specific determination of disease extent compared to 18F-FDG.

Whole body mapping of HER2, an antigen present in multiple cancer types, might (I) Reduce tumor lesion sampling errors and resultingly reduce false negative HER2 IHC outcomes, potentially broadening the therapeutic and interventional treatment options for the patient; (II) Enable identification of inter-and intratumor heterogeneity; and (III) Support follow-up of HER2 targeted treatment response, and accompanied treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years at the time of informed consent signature) male or female patient
2. Patient with confirmed de novo or pre-treated mBC (multiple previous treatment lines in metastatic setting are allowed).
3. Patients with documented hormone receptor positive/HER2 negative, triple-negative or HER2 positive mBC that could become eligible for commercially available HER2 targeted monotherapy (i.e. through confirmation of HER2 IHC non-0 status assessed during the course of the study).
4. Patient presenting with at least one target biopsiable, FDG positive , non-liver metastatic lesion of ≥15 mm defined on ceCT (as part of screening 18F-FDG PET/ceCT assessment).
5. Patient willing to undergo at least one tumor biopsy.
6. Male patients able to father children and female patients of childbearing potential agree to use effective methods of contraception during the diagnostic and SOCa treatment follow-up study phases.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2.
8. Ability and willingness of the research participant to provide written informed consent.

Exclusion Criteria:

1. Primary (non-metastatic) breast cancer.
2. Patient not willing to undergo at least one tumor biopsy. Note: A recent biopsy and accompanied locally assessed IHC/ISH analyses, completed before screening, will not be accepted for study purposes.
3. 18F-FDG PET/ceCT completed before screening and patient not willing to repeat this assessment.
4. Metastatic setting 18F-FDG PET/ceCT indicating that the identified tumor lesions cannot be biopsied due their location and/or tissue type and/or an increased risk for serious comorbidities.
5. Brain and liver metastases are the sole sites of metastatic disease.
6. Life expectancy lower than 3 months.
7. Pregnancy or breastfeeding.
8. Inadequate organ function, suggested by clinically relevant abnormal laboratory results:

   1. Significantly impaired renal function defined as estimated Glomerular Filtration Rate (GFR) <30 ml/min/1.73m2.
   2. Absolute neutrophil count <1,500 cells/mm3.
   3. Total bilirubin ~1.5 x Upper Limit of Normal (ULN) (unless the patient has documented Gilbert's syndrome).
   4. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or Alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SGPT) >5.0 x ULN.
9. Patients with a known hypersensitivity to any of the investigational medicinal product (IMP) components or packaging.
10. Patients with increased risks of bleeding or other complications from biopsies (e.g. patients under anticoagulation therapy for whom temporary discontinuation of this therapy cannot be safely performed).
11. Patients with a known hypersensitivity or contraindication for iodinated contrast media (iCM) which cannot be controlled by taking prophylactic measures (e.g. temporary treatment interruption or introduction of adequate pre-medication).
12. Patients who cannot undergo PET/CT scanning (including but not limited to body size and claustrophobia).
13. Any condition that in the opinion of the investigator may significantly interfere with study compliance (including but not limited to psychological or psychiatric, social or geographical condition potentially hampering compliance with the study requirements).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
positive, negative, and overall diagnostic agreement between 68Ga-ABS011 PET/CT and the standard of care IHC (and ISH) HER2 status test. | immediately after the 68Ga-ABS011 PET/CT procedure
  Evaluation, on a per-lesion level, of the diagnostic performance (positive, negative, and overall diagnostic agreement compiled of ratios between true positive, true negative, false psoitive and false negative 68Ga-ABS011 PET/CT results)) of 68Ga-ABS011 PET/CT(III) compared to HER2 IHC (and ISH) status.

SECONDARY OUTCOMES:
Safety of 68Ga-ABS011. | up to 6 weeks after initiation of the HER2 targeted monotherapy
  Incidence rate of all adverse events (AEs) and serious AEs (SAEs)
Change in treatment management | immediately after the 68Ga-ABS011 PET/CT procedure
  Proportion of patients for whom the whole body 68Ga-ABS011 PET/CT guided biopsy impacted the management of the mBC
reliability of whole body 68Ga-ABS011 PET/CT compared to HER2-targeted treatment response (Early tumor shrinkage) | 6 weeks after initiation of the HER2 targeted monotherapy
  Positive and negative predictive value and likelihood ratio of 68Ga-ABS011 using 18F-FDG PET/ceCT as a reference.
reliability of whole body 68Ga-ABS011 PET/CT compared to HER2-targeted treatment response (metabolic response) | 6 weeks after initiation of the HER2 targeted monotherapy
  Positive and negative predictive value and likelihood ratio of 68Ga-ABS011 using 18F-FDG PET/ceCT as a reference.
Tumor heterogeneity | immediately after the 68Ga-ABS011 PET/CT procedure
  Inter-tumor heterogeneity assessment by measuring the proportion of discordance between the total number of lesions and number of overlapping lesions confirmed on 18F-FDG and/or 68Ga-ABS011 PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Gebhart, Principal Investigator — Institut Jules Bordet Brussels; Evandro De Azambuja, Principal Investigator — Institut Jules Bordet Brussels
Locations (6):
- Belgium (6):
  - OLV Aalst, Aalst, East-Flanders
  - AZ Delta CHIREC, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Free University Brussels (VUB), Brussels
  - Institut Jules Bordet, Brussels
  - University Hospital Gasthuisberg, Leuven

REFERENCES:
- See also: Website Sponsor — https://abscint.com/